CLINICAL TRIAL: NCT07388394
Title: Describe and Evaluate the Impact of Polypharmacy on Healthy Aging in People Living With HIV Over the Age of 75 Who Are Being Treated at Nice University Hospital.
Brief Title: Polypharmacy on Healthy Aging in People Living With HIV Over the Age of 75
Acronym: POLYVIH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25-PP-19
Record Dates: First submitted 2026-01-19; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Virus-HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- people living with HIV over the age of 75 (Other)
  Interventions: Other: interview with advanced practice nurse

INTERVENTIONS:
Other: interview with advanced practice nurse — 45 to 60 minutes of interview

SUMMARY:
Since the advent of antiretroviral treatments, the life expectancy of people living with HIV (PLHIV) has increased significantly. In France, more than 30% of PLHIV are now over 50 years old. This population is exposed to high multimorbidity, leading to frequent polypharmacy, defined as the regular use of at least five medications. Polypharmacy also has a qualitative dimension, including potentially inappropriate prescriptions. It increases the risk of adverse effects and drug interactions and impairs quality of life. A coordinated geriatric approach is therefore essential to optimize care. Healthy aging, promoted by the WHO, aims to improve the lives of older people. In this context, a study will be conducted at the Nice University Hospital among PLHIV aged 75 and over. It will collect quantitative data, the results of which will enable us to consider, if necessary, adapting the care pathways of these patients whose needs are complex.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Aged 75 or over
* Affiliated with the social security system
* Having expressed no objection to participating in the study

Exclusion Criteria:

* Refusal to participate
* Known severe cognitive impairment preventing the interview from being conducted
* Patient under guardianship or conservatorship

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Describe polypharmacy among people living with HIV aged 75 and older. | 15 months
  The average number of medications taken

SECONDARY OUTCOMES:
Assess the most common comorbidities associated with polypharmacy in the population of PLHIV aged 75 | 15 months
  Number et type of comorbidities
Assess whether people taking multiple medications have a lower treatment adherence score than those taking fewer medications. | 15 months
  Score obtained on the Morisky MMAS-8 questionnaire
Assess the level of functional independence in this age group and link it to the existence of polypharmacy. | 15 months
  Lawton and Brody IADL scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, CHU de Nice, France

IPD SHARING:
Plan to Share IPD: No